CLINICAL TRIAL: NCT06765109
Title: A Phase 3 Study of the Selective Anaplastic Lymphoma Kinase (ALK) Inhibitor NVL-655 Compared to Alectinib in First-Line Treatment of Patients With ALK-Positive Advanced Non-Small Cell Lung Cancer (ALKAZAR)
Brief Title: Neladalkib (NVL-655) for TKI-naive Patients With Advanced ALK-Positive NSCLC
Acronym: ALKAZAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nuvalent Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NVL-655-04; 2024-517553-26 (EudraCT Number)
Expanded Access: NCT06834074 (Available)
Record Dates: First submitted 2024-11-08; First posted 2025-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer; Anaplastic Lymphoma Kinase-positive
Keywords: NSCLC; Lung cancer; Lung neoplasms; Lung diseases; ALK positive NSCLC; TKI naive; ALK TKI naive; Treatment naive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Lung Diseases | interventions — alectinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neladalkib (NVL-655) (Experimental): 150mg taken orally once daily (QD)
  Interventions: Drug: Neladalkib (NVL-655)
- Alectinib (Active Comparator): 600mg taken orally twice daily (BID)
  Interventions: Drug: Alectinib

INTERVENTIONS:
Drug: Neladalkib (NVL-655) — Oral tablet of Neladalkib (NVL-655)
  Arms: Neladalkib (NVL-655)
Drug: Alectinib — Oral capsule of alectinib
  Other Names: Alecensa
  Arms: Alectinib

SUMMARY:
Multicenter, randomized, controlled, open-label, Phase 3 study designed to demonstrate that neladalkib (NVL-655) is superior to alectinib in prolonging progression-free survival (PFS) in patients with treatment-naïve, Anaplastic Lymphoma Kinase (ALK) positive, advanced Non-Small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 ratio (approximately 225 in each arm) to receive either neladalkib (NVL-655) or alectinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced (not amenable for multimodality treatment) or metastatic Non-small Cell Lung Cancer (NSCLC)
2. Documented Anaplastic Lymphoma Kinase (ALK) rearrangement via testing of tissue or blood
3. No prior systemic anticancer treatment for NSCLC (adjuvant/neoadjuvant chemotherapy allowed if 12 months prior to randomization; prior ALK tyrosine kinase inhibitor [TKI] such as alectinib is not allowed in any setting)
4. Measurable disease (1 or more target lesions per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
5. Pretreatment tumor tissue

Exclusion Criteria:

1. Patient's cancer has a known oncogenic driver alteration other than ALK.
2. Known allergy/hypersensitivity to excipients of neladalkib or alectinib.
3. Ongoing or recent radiotherapy as per protocol-specified timeframes prior to randomization
4. Major surgery within 4 weeks prior to randomization
5. Uncontrolled clinically relevant infection requiring systemic therapy
6. Known active tuberculosis, or active Hepatitis B or C
7. QT corrected for heart rate by Fridericia's formula (QTcF) > 470 msec on repeated assessments
8. Clinically significant cardiovascular disease
9. Brain metastases associated with progressive neurological symptoms or requiring increasing doses of corticosteroids to control CNS disease
10. Active malignancy requiring therapy within 2 years prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) per blinded independent central review (BICR) | Up to 5 years after first patient dosed
  Time from randomization to BICR-assessed radiographic disease progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years after first patient dosed
  Time from randomization to death
Progression-free survival (PFS) per investigator assessment | Up to 5 years after first patient dosed
  Time from randomization to investigator-assessed radiographic disease progression or death
Time to intracranial progression per BICR | Up to 5 years after first patient dosed
  Time from randomization to the first BICR-assessed occurrence of disease progression in the central nervous system (CNS)
Intracranial objective response rate (IC-ORR) | Up to 5 years after first patient dosed
  Proportion of patients with a confirmed intracranial response (intracranial complete response [IC-CR] or intracranial partial response [IC-PR]) among patients with measurable CNS disease at baseline
Intracranial duration of response (IC-DOR) | Up to 5 years after first patient dosed
  Time from first intracranial response (IC-CR or IC-PR) to radiographic intracranial disease progression or death
Objective response rate (ORR) | Up to 5 years after first patient dosed
  Proportion of patients with a complete response or partial response
Duration of response (DOR) | Up to 5 years after first patient dosed
  Time from first response (complete or partial) to radiographic disease progression or death
Intracranial progression per investigator assessment | Up to 5 years after first patient dosed
  Time to investigator-assessed intracranial progression
Treatment-emergent adverse events (TEAEs) and changes in clinically relevant laboratory parameters | Up to 5 years after first patient dosed
  Incidence and severity of TEAEs and changes in clinically relevant laboratory parameters
Patient-reported measures in health-related quality of life (QoL) | Up to 5 years after first patient dosed
  Changes in patient-reported outcomes (PROs) assessed by the European Organization for Research and Treatment of Cancer QoL core questionnaire - Cancer (EORTC QLQ-C30)
Patient-reported measures in lung cancer symptoms and side effects of treatment | Up to 5 years after first patient dosed
  Changes in PROs assessed by the European Organization for Research and Treatment of Cancer QoL - Lung Cancer module (EORTC QLQ-LC29)
Patient-reported measures in patient functioning | Up to 5 years after first patient dosed
  Changes in PROs assessed by the European Quality of Life (EuroQol) 5-dimension questionnaire (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Viola Zhu, MD, PhD, Study Director — Nuvalent Inc.
Locations (98):
- United States (17):
  - Palo Verde Hematology Oncology, Glendale, Arizona
  - University of California, Irvine Health, Orange, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Sylvester Comprehensive Cancer Center Miami, Miami, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University Center for Advanced Medicine, St Louis, Missouri
  - Clinical Research Alliance Inc., New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
- Argentina (2):
  - Sanatorio Parque S.A., Rosario, Santa Fe Province
  - Sanatorio Allende, Córdoba
- Australia (2):
  - Westmead Hospital, Westmead, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
- A.C.Camargo Cancer Center, São Paulo, Brazil
- Nemocnice AGEL Nový Jičín a.s., Nový Jičín, Czechia
- Denmark (2):
  - Herlev and Gentofte Hospital, Herlev
  - University of Southern Denmark, Odense
- France (9):
  - Centre Hospitalier Universitaire d' Angers, Angers
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Leon Berard, Lyon
  - Hospital Nord, Marseille
  - Institut Regional du Cancer de Montpellier, Montpellier
  - Centre Hospitalier Universitaire (CHU) Nantes Hopital Nord Laennec, Nantes
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Pessac
  - Centre Hospitalier Universitaire de Toulouse - Hopital Larrey, Toulouse
- Germany (3):
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - LungenClinic Grosshansdorf GmBH, Großhansdorf
  - Lungenfachklinik Immenhausen, Immenhausen
- Greece (5):
  - Henry Dunant Hospital Center, Athens
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - University General Hospital of Larissa, Larissa
  - Athens Medical Center, Marousi
  - Bioclinic Thessaloniki, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital Department of Medicine, Hong Kong
  - Prince of Wales Hospital, Shatin
- Matrai Gyogyintezet, Gyöngyös, Hungary
- Italy (4):
  - Azienda Ospedaliero Universitaria delle Marche, Ancona
  - Istituto Clinico Humanitas, Milan
  - AUSL Della Romagna - Ospedale Santa Maria delle Croci, Ravenna
  - Istituti Fisioterapici Ospitalieri - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
- Japan (3):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Malaysia (5):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Institut Kanser Negara, Putrajaya, Putrajaya
  - Beacon International Specialist Centre, Petaling Jaya, Selangor
  - Hospital Umum Sarawak, Kuching
- Netherlands (2):
  - Nederlands Kanker Instituut-Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - University Medical Center Utrecht, Utrecht
- Poland (3):
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - One Day Med, Szczecin
- Portugal (4):
  - Hospital de Cascais, Alcabideche
  - Fundacao Champalimaud, Lisbon
  - CUF Porto Hospital, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E., Porto
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Center for Lung Cancer, National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei Cancer Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Complejo Hospitalario Universitario a Coruña, A Coruña
  - UOMi Cancer Center, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (4):
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- United Kingdom (7):
  - Cambridge University Hospitals NHS Trust, Addenbrooke's Hospital, Cambridge
  - Royal Free London NHS Foundation Trust, Hampstead
  - Guy's Cancer Centre NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Maidstone Hospital, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham City Hospital, Nottingham